CLINICAL TRIAL: NCT04717895
Title: Psychological and Postural Effects of Exposure to Both Types of Virtual Environments
Acronym: PREUV
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Gérond'if (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 2020-A01999-30
Record Dates: First submitted 2020-12-18; First posted 2021-01-22 (Actual); Last update posted 2023-01-17 (Actual); Status verified 2023-01

CONDITIONS: Autonomous Subjects, Aged 65 and Afraid of Falling
Keywords: Fear of falling; Postural changes; Stand upright without technical assistance

STUDY DESIGN:
Intervention Model Description: Randomization will be carried out after inclusion and allocation of a selection / inclusion number of subjects and will be carried out as follows:
  * Subjects included and who will be identified with an even selection number will begin the virtual reality session by viewing a rocking environment followed by a translation environment
  * Subjects included and who will be identified with an odd selection number will start the virtual reality session by viewing a translation environment followed by a rocking environment
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- 1st Situation (Experimental): Subjects included will be identified with an even selection number will begin the virtual reality session by viewing a rocking environment followed by a translation environment
  Interventions: Diagnostic Test: Rocking environment forward (B) followed by a translation environment
- 2nd Situation (Active Comparator): Subjects included will be identified with an odd selection number will start the virtual reality session by viewing a translation environment followed by a rocking environment
  Interventions: Diagnostic Test: Translation environment followed by a rocking environment

INTERVENTIONS:
Diagnostic Test: Rocking environment forward (B) followed by a translation environment — Start by the virtual reality session by viewing a rocking environment followed by a translation environment
  Arms: 1st Situation
Diagnostic Test: Translation environment followed by a rocking environment — Start by the virtual reality session by viewing a translation environment followed by a rocking environment
  Arms: 2nd Situation

SUMMARY:
The main aim of this study is to compare the fear of falling induced by each type of virtual scene (rocking and translation). Fear of falling will be assessed by a numerical fear of falling scale.

The benefits for the participants would be the discovery of Virtuel Reality, the awareness of their fear of falling and its repercussions on posture and, if necessary, referral to specialized rehabilitation centers. This study will provide evidence on the context of the emergence of the fear of falling in order to propose, in perspective, appropriate rehabilitation management procedures.

DETAILED DESCRIPTION:
This bicentric study will proceed as follows:

* Complete clinical examination, carried out as part of your consultation in a day hospital.
* Perform a virtual reality session of about 2 hours. This session will take place as follows:

  * Wear a virtual reality headset. The helmet is compatible with the wearing of glasses.
  * View a virtual scene for two minutes in order to familiarize yourself with the device. This first viewing will be followed by a 10 minute break.
  * Then the patient will be placed on a rectangular platform (Wii Balance Board - WBB)
  * Give the virtual reality headset again to the patient, who will view a 2-minute series of a series of 2 minutes in a standing position comprising a moving virtual environment (one tilting forward and another in forward translation).
  * After a 10 minute break, the session will continue with 4 other sets of 5 minutes duration (5 times 1 minute of a forward tilt or forward translation scene). These 4 series will be separated by 10 min break
  * During each break, the patient participating in the study will complete a questionnaire on the possible side effects of virtual reality (cybermalaise).

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 65 years old
* Declaring to be able to maintain the upright station without technical assistance for at least 5 minutes
* Being afraid of falling with a score greater than or equal to 23 on the Falls Efficacy Scale-International questionnaire (Yardley et al., 2005)
* Good understanding of the French language
* Benefiting from a social security system
* Have read the information notice and have consented to participate in the study by signing a written consent

Exclusion Criteria:

* Severe cognitive impairment according to DMS-5 criteria
* Medical diagnosis of neurological disease
* Trauma dating less than 6 months to the lower limb
* Symptoms of vestibular or cerebellar involvement
* Major visual disorder defined by visual acuity of one or both eyes less than or equal to 3 / 10th without correction
* History of epileptic seizure: this is a total contraindication due to proximity to a screen (Virtual Reality Ethics Committee, 2019)
* Psychiatric disorders (Schizophrenia, dissociative disorders, borderline state, paranoia)

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 44 (Estimated)
Dates: Start 2022-04-24 (Actual); Primary Completion 2023-10 (Estimated); Study Completion 2024-02 (Estimated)

PRIMARY OUTCOMES:
measurement of fear of falling using a Numeric scale of fear of falling | 2 Hours

SECONDARY OUTCOMES:
assess posture by recording the coordinates of center of pressure during exposure to Virtual Reality using the Wii Balance Board (WBB) | 2 Hours
Evaluate the subjective perception of stability which will be evaluated using a numerical scale of the perception of stability | 2 Hours
Cyber sickness will be assessed by the Simulator Sickness Questionnaire | 2 Hours

CONTACTS AND LOCATIONS:
Overall Officials: Emmanuelle DURON, MD, Study Chair — Geriatric Department, Paul Brousse Hospital
Locations (1):
- Geriatric Department, Paul Brousse Hospital, Villejuif, Île-de-France Region, France